CLINICAL TRIAL: NCT05834491
Title: A Novel Approach to Plantar Fasciitis in the Aging Population
Acronym: NAPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: University of Hartford (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Irene Davis, Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY004876; 1R01AG071646 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-04-28 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Plantar Fasciitis, Chronic
Keywords: minimal footwear, pain, function, strengthening
MeSH Terms: conditions — Fasciitis, Plantar; Pain | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Footwear (Vivobarefoot) (Experimental): The experimental intervention involves the combination of foot strengthening/stretching and minimal footwear to promote the foot strengthening beyond the exercise program to mitigate weakening from chronic support.
  Interventions: Device: minimal shoes and foot strengthening and flexibility exercises
- Supportive Footwear (Active Comparator): The control intervention is considered the standard of care and involves combination of foot stretching and the addition of supportive shoes and foot orthoses.
  Interventions: Device: Supportive Footwear, foot orthotic device and foot flexibility exercises

INTERVENTIONS:
Device: minimal shoes and foot strengthening and flexibility exercises — Flexible shoes that do not provide support and exercises aimed at increasing the strength of plantar intrinsic and extrinsic foot muscles along with foot flexibility exercises aimed at increasing the range of motion of the foot and ankle
  Arms: Minimal Footwear (Vivobarefoot)
Device: Supportive Footwear, foot orthotic device and foot flexibility exercises — sturdy supportive shoes fitted with supportive foot orthotic devices and foot flexibility exercises aimed at increasing the range of motion of the foot and ankle
  Arms: Supportive Footwear

SUMMARY:
The goal of this study is to determine whether improving foot strength through foot exercises and minimal footwear can provide improved outcomes over the short and long term. The main research question it aims to answer is: Can the minimal footwear intervention be used to improve the health of aging adults with plantar fasciitis?? Participants will be randomized into 2 groups. One group will receive minimal shoes and foot strengthening and foot flexibility exercises. The other group will receive supportive shoes, foot orthotic device and foot flexibility exercises. Participants' step count will also be monitored.

Researchers will compare pain and physical function between the minimal footwear (MF) and the foot orthotic (FO) groups at each of the follow-up sessions.

DETAILED DESCRIPTION:
Twenty five percent of older adults experience foot pain. Plantar fasciitis, a repetitive strain injury, is one of the most common causes of foot pain in this population. Ten percent of aging adults experience plantar fasciitis with 50% of the cases being disabling. Foot pain can lead to other problems such as reduced mobility, depression and prescription medication use, leading to a reduced quality of life. Foot pain has been related to foot weakness, reduced static and dynamic balance, and reduced walking speed in aging adults.

The standard of care for plantar fasciitis is to brace the arch with foot orthoses and supportive shoes, thereby reducing the strain on the plantar fascia. However, arch support has been shown to be an ineffective long-term strategy for reducing foot pain, as well as leading to intrinsic foot muscle atrophy. As plantar fasciitis is associated with this atrophy, treating it with chronic arch support only increases the risk for recurrence. In fact, there is a 50% recurrence rate and a 45.6% risk of having plantar fasciitis 10 years after the onset of symptoms, and this risk increases with age.

Minimal shoes are designed to allow the foot to function naturally, as if barefoot, which have already been successfully implemented in older adults for the treatment of knee osteoarthritis. Minimal shoes are highly flexible and lack the support of conventional footwear. This places a greater demand on the foot muscles, which promotes strengthening. Indeed, studies of gradual transitioning to walking in minimal shoes have demonstrated significant increases in intrinsic foot muscle size and strength. Stronger foot intrinsic foot muscles have been shown to reduce the strain on the plantar fascia with each step, thereby reducing the risk of developing plantar fasciitis. This is especially important in the older population who develop muscle weakness as they age.

The overall objective of this study is to improve treatment interventions for plantar fasciitis in aging adults. The central hypothesis of this research is that strong intrinsic foot muscles will reduce the strain on the plantar fascia. This, in turn will result in resolution of pain, with less recurrence of plantar fasciitis than the standard of care. The investigators will test this hypothesis by comparing an intervention of stretching, foot orthoses and supportive shoes to one of foot stretching, strengthening and transition to minimal footwear. Training the foot of a patient with plantar fasciitis to function with less support is a significant paradigm shift from interventions aimed at passively supporting the foot. However, the investigators hypothesize that the dynamic stability of the foot muscles will be more effective than a static foot orthosis, that has been shown to promote foot weakening. The investigators will assess outcomes of foot pain, functional activities, and muscle strength, size and function at the 3- and 6-month follow-up, and the incidence of recurrence of plantar fasciitis at the 12 month time point.

ELIGIBILITY:
Inclusion Criteria:

1 Active plantar fasciitis for a minimum of 6 months. 2. Heel/arch pain on first step in the morning, 3. Heel/arch pain with prolonged standing (>15 min), 4. Heel/arch pain with prolonged walking (>15 min), 5. Be able to stand and walk for 10 minutes with little or no pain (<3/10 on a NRPS).

Exclusion Criteria:

1. Having systemic disease such as diabetes, gout, arthritis, neuropathy, surgical reconstructions
2. Having a history of heel surgery or had a steroid injection for heel pain in the past 6 months.
3. Used foot orthoses less than 3 months before start date of study.
4. Having used minimal shoes at any time in the past.
5. No special or vulnerable populations will be recruited.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will testing biomechanical changes which is depends on the gender that they were born. Therefore, eligibility will not be based on their self-representative identification
Enrollment: 138 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Foot Health Status Questionnaire (FHSQ) | Baseline
  It is a self-report questionnaire that relies on participant recall over the previous 7 days. The FHSQ incorporates questions that address foot pain, function, footwear, and general health and activity levels. It is ranged from 1 to 100, where 0 indicates poor foot health and 100 is excellent foot health score. High reliability and validity have been established for it.
Foot Health Status Questionnaire (FHSQ) | 3 months
  It is a self-report questionnaire that relies on participant recall over the previous 7 days. The FHSQ incorporates questions that address foot pain, function, footwear, and general health and activity levels. It is ranged from 1 to 100, where 0 indicates poor foot health and 100 is excellent foot health score. High reliability and validity have been established for it.
Foot Health Status Questionnaire (FHSQ) | 6 months
  It is a self-report questionnaire that relies on participant recall over the previous 7 days. The FHSQ incorporates questions that address foot pain, function, footwear, and general health and activity levels. It is ranged from 1 to 100, where 0 indicates poor foot health and 100 is excellent foot health score. High reliability and validity have been established for it.
Foot pain | Baseline
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 1 month
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 2 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 3 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 4 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 5 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 6 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 7 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 8 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 9 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 10 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 11 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Foot pain | 12 months
  Over the past 7 days on a Numerical Pain Rating Scale from 0 -10 (with 0 being no pain and 10 being the worst pain imaginable) will be asked to participants. The average of weekly pain will be calculated for each months. The questions are as below;
  1. What is the worst your pain has been upon first step in the morning.
  2. What is the worst your pain has been during the day.
  3. Do you have any other foot or lower extremity pain that is limiting your walking?
Step counts | Baseline
  Over the past 7 days of step counts will be monitored via Garmin watch. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 1 month
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 2 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 3 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 4 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 5 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 6 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 7 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 8 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 9 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 10 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 11 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Step counts | 12 months
  Over the past 7 days of step counts will be monitored via Garmin watch. The average of weekly step counts will be calculated for each months. The Garmin watch device was chosen as it has a 1 yr battery life eliminating the need for recharging and is waterproof. It can store 30 days worth of data and also syncs to an app on the participant's smart phone or computer. Therefore, we can access the data directly, eliminating the need for the participants to keep track of their data.
Global Rating Outcome Change (GROC) | 3 months
  GRC scale asks that a person assess his or her current health status, recall that status at a previous time-point. The question is as below.
  With respect to you previous pain, how would you describe yourself now?
Global Rating Outcome Change (GROC) | 6 months
  GROC scale asks that a person assess his or her current health status, recall that status at a previous time-point. The question is as below.
  With respect to you previous pain, how would you describe yourself now?
Patient Acceptable Symptom State (PASS) | 3 months
  This is a single assessment self-reported tool. The question is as below. Taking into account your previous pain status, do you consider your foot health satisfactory?
Patient Acceptable Symptom State (PASS) | 6 months
  This is a single assessment self-reported tool. The question is as below. Taking into account your previous pain status, do you consider your foot health satisfactory?

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Baseline
  It is a self-report questionnaire that quantifies physical activity over the previous 7 days. It includes questions specific to time spent walking, as well as sedentary behavior such as time spent sitting. The scale of IPAQ is between 500 -10000 MET. High reliability and validity have been established for it.
International Physical Activity Questionnaire (IPAQ) | 3 months
  It is a self-report questionnaire that quantifies physical activity over the previous 7 days. It includes questions specific to time spent walking, as well as sedentary behavior such as time spent sitting. The scale of IPAQ is between 500 -10000 MET. High reliability and validity have been established for it.
International Physical Activity Questionnaire (IPAQ) | 6 months
  It is a self-report questionnaire that quantifies physical activity over the previous 7 days. It includes questions specific to time spent walking, as well as sedentary behavior such as time spent sitting. The scale of IPAQ is between 500 -10000 MET. High reliability and validity have been established for it.
Static and dynamic balance | Baseline
  This test has been used as a measure of physical performance in older adults. Participants will stand, barefoot and on one leg, on a force plate that is at the center of a grid marked by 3 pieces of tape. They will perform maximal reaches with the non-supporting leg along each of the taped lines (Anterior, Posterior-Lateral, and Posterior-Medial). The maximum distance they reached will be measured in centimeter.
Static and dynamic balance | 3 months
  This test has been used as a measure of physical performance in older adults. Participants will stand, barefoot and on one leg, on a force plate that is at the center of a grid marked by 3 pieces of tape. They will perform maximal reaches with the non-supporting leg along each of the taped lines (Anterior, Posterior-Lateral, and Posterior-Medial). The maximum distance they reached will be measured in centimeter.
Static and dynamic balance | 6 months
  This test has been used as a measure of physical performance in older adults. Participants will stand, barefoot and on one leg, on a force plate that is at the center of a grid marked by 3 pieces of tape. They will perform maximal reaches with the non-supporting leg along each of the taped lines (Anterior, Posterior-Lateral, and Posterior-Medial). The maximum distance they reached will be measured in centimeter.
Muscles size of cross sectional area | Baseline
  It will be measured with ultrasound imaging. These muscles are the flexor digitorum brevis (FDB), abductor hallicus (ABDH), abductor digiti minimi (ADM) and quadratus plantae (QP). The ultrasound probe (GE Logiq S8, 6-15Mhz linear array) with gel will be placed in alignment with internal bony landmarks (e.g. metatarsal head and navicular tuberosity) or external landmarks (e.g. 30% and 50% of leg length from knee joint line marked on the skin surface) to standardize measurement location.
Muscles size of cross sectional area | 3 months
  It will be measured with ultrasound imaging. These muscles are the flexor digitorum brevis (FDB), abductor hallicus (ABDH), abductor digiti minimi (ADM) and quadratus plantae (QP). The ultrasound probe (GE Logiq S8, 6-15Mhz linear array) with gel will be placed in alignment with internal bony landmarks (e.g. metatarsal head and navicular tuberosity) or external landmarks (e.g. 30% and 50% of leg length from knee joint line marked on the skin surface) to standardize measurement location.
Muscles size of cross sectional area | 6 months
  It will be measured with ultrasound imaging. These muscles are the flexor digitorum brevis (FDB), abductor hallicus (ABDH), abductor digiti minimi (ADM) and quadratus plantae (QP). The ultrasound probe (GE Logiq S8, 6-15Mhz linear array) with gel will be placed in alignment with internal bony landmarks (e.g. metatarsal head and navicular tuberosity) or external landmarks (e.g. 30% and 50% of leg length from knee joint line marked on the skin surface) to standardize measurement location.
Muscle Strength | Baseline
  Strength of the intrinsic muscles will be measured with a force dynamometer.
Muscle Strength | 3 months
  Strength of the intrinsic muscles will be measured with a force dynamometer.
Muscle Strength | 6 months
  Strength of the intrinsic muscles will be measured with a force dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Flroida, Tampa, Florida, United States